CLINICAL TRIAL: NCT02127788
Title: Observational, Longitudinal, Prospective, French, Multicentre Study Conducted on Adult and Paediatric Patients Treated With Micafungin in Prophylaxis and Followed Over a 3 Months' Period in Routine Medical Practice
Brief Title: Use of Micafungin (Mycamine®) as Antifungal Prophylaxis in Haematology and Onco-haematology
Acronym: OLYMPE
Status: Completed | Type: Observational
Sponsor: Astellas Pharma S.A.S. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: FR-MYC-NI-003
Record Dates: First submitted 2014-04-17; First posted 2014-05-01 (Estimated); Last update posted 2024-10-21 (Actual); Status verified 2019-03

CONDITIONS: Antifungal Prophylaxis; Haemopathy
Keywords: Haematology; Micafungin; Observational study; Prophylaxis; Invasive Fungal Infection; France
MeSH Terms: conditions — Invasive Fungal Infections | interventions — Micafungin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Micafungin: Patients affected with haemopathy (or affected with solid tumor for paediatric patients) under antifungal prophylaxis with micafungin.
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — intravenous
  Other Names: FK463; Mycamine

SUMMARY:
The purpose of this observational study is to describe the actual conditions of prescription of micafungin in antifungal prophylaxis in French haematological and onco-haematological units. The efficacy and the safety outcomes will be described.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with haemopathy or paediatric patients with haemopathy or solid tumor.
* Patient hospitalized in haematology, onco-haematology or onco-paediatrics unit.
* Patient initiating antifungal prophylaxis with micafungin.

Exclusion Criteria:

* Patient presenting documented fungal infection.
* Patient already included in a biomedical study impacting the care management of invasive fungal infection at the time of inclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized, adult patients with haemopathy or paediatric patients with haemopathy or solid tumor, under antifungal prophylaxis with micafungin.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-07-03 (Actual); Primary Completion 2016-01-27 (Actual); Study Completion 2016-01-27 (Actual)

PRIMARY OUTCOMES:
Breakthrough incidence of Invasive Fungal Infection (IFI), defined according to the revised EORTC/MSG criteria, during prophylaxis use of micafungin | Up to 3 months
  EORTC/MSG : European Organization for Research and Treatment of Cancer/ Invasive Fungal Infections Cooperative Group and the National Institute of Allergy and Infectious Diseases Mycoses Study Group

SECONDARY OUTCOMES:
Odds ratio and 95% CI for each identified risk factors | Up to 3 months
Incidence of IFI, defined according to the revised EORTC/MSG criteria | Up to 3 months
Characteristics of patients treated with micafungin | Day 0 (start of prophylaxis)
Conditions of use of micafungin | Up to 3 months
  dose and administration pattern, temporary interruptions and treatment duration, oral treatment take-over
Description of adverse events (AE) and serious adverse events (SAE) | Up to 3 months
Characteristics of units | Day 0
  participating physicians (age, status, specialty), type of institution, location , type of unit, size of unit

CONTACTS AND LOCATIONS:
Overall Officials: Medical and Scientific Affairs Manager, Infectious Diseases, Study Director — Astellas Pharma S.A.S.
Locations (14):
- France (14):
  - Site, Angers
  - Site, Béziers
  - Site, Bordeaux
  - Site, Brest
  - Site, Clermont-Ferrand
  - Site, Lille
  - Site, Limoges
  - Site, Marseille
  - Site, Metz
  - Site, Montpellier
  - Site, Nantes
  - Site, Paris
  - Site, Saint-Denis La Réunion
  - Site, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.